CLINICAL TRIAL: NCT05474209
Title: The Combined Impact of a Structured Tai Chi Exercise Program on Selected Clinical Aspects and Quality of Life of Patients With Multiple Sclerosis
Brief Title: Effect of Tai Chi on Balance, Mood, Cognition, and Quality of Life in Patients With Multiple Sclerosis
Acronym: TaiChi-SM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC/0130/2020/UNBKramare
Record Dates: First submitted 2022-06-16; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Tai Chi Chuan; balance; non-pharmacological interventions; physical therapy; posturography
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The intervention study will include treated patients with relapsing-remitting MS who meet the 2010 MR McDonald criteria for dissemination in time and space, last month before enrollment without relapse, no severe cognitive impairment, and according to the Kurtz Disability Scale (EDSS). 4.5 for 12 months and exercise intensity three times a week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise patients with multiple sclerosis (Active Comparator): a group that undergoes a "tai-chi" intervention - a special program for patients with multiple sclerosis - once a week with a Tai Chi instructor lasting 90 minutes. At V0, each patient will receive an accurate instructional video for a separate home exercise "tai-chi" at an intensity of twice a week.
  Interventions: Other: "Tai-chi" - a special program for patients with multiple sclerosis - once a week training with a Tai Chi instructor lasting 90 minutes
- non-exercising patients with multiple sclerosis (No Intervention): the group will be a control group, patients with multiple sclerosis undergo a whole battery of examinations and scales, they will not undergo exercise.

INTERVENTIONS:
Other: "Tai-chi" - a special program for patients with multiple sclerosis - once a week training with a Tai Chi instructor lasting 90 minutes — "Tai-chi" - a special program for patients with multiple sclerosis - once a week training with a Tai Chi instructor lasting 90 minutes for 12 months
  Arms: exercise patients with multiple sclerosis

SUMMARY:
Multiple sclerosis (MS) is an inflammatory and neurodegenerative disease of the central nervous system (CNS). The clinical picture is very variable, ultimately resulting in disability. Disease attacks manifest themselves depending on the location of the CNS damaged by inflammation, demyelination, axonal loss and gliosis. The most common manifestations include motor disorders with the development of stiffness, balance and coordination, cognition, fatigue and depression. In the long term, most patients with MS will achieve significant and irreversible incapacitation. Immunomodulatory therapy is designed to reduce disease activity, slowing progression, but only to a certain extent. A significant benefit, but little researched, is physical exercise. Tai Chi has a positive effect on various neurological diseases. In recent studies, Tai Chi has shown improvements in coordination and balance, depression, anxiety, cognition and overall quality of life in patients with MS. The aim of the project is to assess the therapeutic value of structured Tai Chi exercise based on published clinical work.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic disease that mainly affects young people with a maximum incidence in working age. Demyelination, axial damage, inflammation and gliosis affect the brain, spinal cord and optic nerves. The resulting symptoms are both physical and mental, and are closely related. The degree of disability in MS can range from relatively benign to malignant forms leading to severe disability in patients over several years. The most common symptoms of MS are impaired motor and sensitive functions, imbalances and coordination. Loss of balance leads to falls, in patients with MS they occur with a prevalence of 34-64%. The result is injuries, fractures, soft tissue damage, restricted activities and reduced mobility. The psychological aspect is loss of independence, social isolation, reduced quality of life. The clinical picture of MS also includes cognitive dysfunction (more than half of patients with MS) and a number of neurobehavioral disorders, especially fatigue (53-90%), depression (with a prevalence of 40-60%), anxiety disorders (35%). They are conditioned not only by reactivity, but indeed by the pathophysiology of the disease itself. Cognitive and affective symptoms associated with MS are a serious psychosocial factor limiting the course of the disease. MS is an incurable disease. Immunomodulatory therapy, which is continuously modified according to the patient's condition, is essentially a variety of effective prevention of progression of disability. At present, there is not enough knowledge about the right combination and structure of programmed physical exercise, which would significantly alleviate the symptoms of MS. While in the past it has not been recommended to patients in the traditional sense of MS, recent findings integrate physical exercise into the treatment of MS as an essential component. Current research points to significant benefits of physical activity in patients with MS: improved aerobic capacity and muscle strength, mobility, fatigue, and quality of life. Even the potential of physical exercise for the pathology of SM itself is expected, namely anti-inflammatory - by modulating the cytokine profile of T-cells and neuroprotective - by increasing the level of serum BDNF (brain-derived neurotrophic factor). Tai Chi Chuan - The inner art of Taoist Tai Chi is not practiced as a martial art technique or in a competitive spirit. A characteristic feature of Tai Chi is stretching and rotation in every movement. Another aspect is the emphasis on sitting and getting up, which helps to improve balance, strengthen legs, tendons and ligaments. Tai Chi also has a spiritual dimension associated with physical exercise. The primary goal is relaxation of body and soul, for Tai Chi are characterized by slow and controlled movements, deep relaxed breathing and correct posture through a state of awareness and concentration. Tai Chi improves flexibility, range of motion, muscle strength and balance and therefore could be beneficial for MS patients. As many of the basic principles of Tai Chi are directly related to postural control, initial smaller studies have begun to show that improvements in depression, quality of life and balance have improved.

ELIGIBILITY:
Inclusion Criteria:

1. clinically defined MS,
2. age from 20 to 60 years,
3. and the ability to stand and walk independently at least 200 meters without an assistive device.

Exclusion Criteria:

1. clinical MS exacerbation during the study,
2. disease-modifying drug change during the study,
3. pregnancy,
4. involvement in any other exercise programme,
5. severe cognitive deficit (defined by Montreal Cognitive Assessment score ≤19), and
6. any other health condition that would interfere with an exercise programme (such as musculoskeletal disorder, lung, or heart disease).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
V0 visit- Static posturography | 1. day
  Static posturography- eyes closed on the foam rubber in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V1 visit- Static posturography | 3 months after V0 visit
  Static posturography- eyes closed on the foam rubber in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V2 visit- Static posturography | 6 months after V0 visit
  Static posturography- eyes closed on the foam rubber in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V3 visit- Static posturography | 9 months after V0 visit
  Static posturography- eyes closed on the foam rubber in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V4 visit- Static posturography | 12 months after V0 visit
  Static posturography- eyes closed on the foam rubber in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V0 visit- Static posturography LI | 1. day
  Static posturography- - LI - line integral in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V1 visit- Static posturography LI | 3 months after V0 visit
  Static posturography- - LI - line integral in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V2 visit- Static posturography LI | 6 months after V0 visit
  Static posturography- - LI - line integral in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V3 visit- Static posturography LI | 9 months after V0 visit
  Static posturography- - LI - line integral in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V4 visit- Static posturography LI | 12 months after V0 visit
  Static posturography- - LI - line integral in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V0 visit- Static posturography TA | 1. day
  Static posturography- TA - total area in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V1 visit- Static posturography TA | 3 months after V0 visit
  Static posturography- TA - total area in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V2 visit- Static posturography TA | 6 months after V0 visit
  Static posturography- TA - total area in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V3 visit- Static posturography TA | 9 months after V0 visit
  Static posturography- TA - total area in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V4 visit- Static posturography TA | 12 months after V0 visit
  Static posturography- TA - total area in mm2, Objective test (instrumental), Score interpretation: The more, the worse.
V0 visit- Static posturography RMS | 1. day
  Static posturography- - RMS - root mean square in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V1 visit- Static posturography RMS | 3 months after V0 visit
  Static posturography- - RMS - root mean square in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V2 visit- Static posturography RMS | 6 months after V0 visit
  Static posturography- - RMS - root mean square in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V3 visit- Static posturography RMS | 9 months after V0 visit
  Static posturography- - RMS - root mean square in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V4 visit- Static posturography RMS | 12 months after V0 visit
  Static posturography- - RMS - root mean square in mm, Objective test (instrumental), Score interpretation: The more, the worse.
V0 visit- Mini-BESTest | 1. day
  Mini-BESTest - Balance Evaluation Systems Test measure in points from 0 - 28. Objective test (clinical), The less, the worse.
  The Mini-BESTest consists of 14 tasks that assess static, proactive, and reactive balance. This balance measure is a shorter version of the original 27-item BESTest and takes only 15 minutes to administer. The mini-BESTest may be more appropriate and effective for ambulatory people with MS with relatively few walking disabilities. Higher scores mean better outcome.
V1 visit- Mini-BESTest | 3 months after V0 visit
  Mini-BESTest - Balance Evaluation Systems Test measure in points from 0 - 28. Objective test (clinical), The less, the worse.
  The Mini-BESTest consists of 14 tasks that assess static, proactive, and reactive balance. This balance measure is a shorter version of the original 27-item BESTest and takes only 15 minutes to administer. The mini-BESTest may be more appropriate and effective for ambulatory people with MS with relatively few walking disabilities. Higher scores mean better outcome.
V2 visit- Mini-BESTest | 6 months after V0 visit
  Mini-BESTest - Balance Evaluation Systems Test measure in points from 0 - 28. Objective test (clinical), The less, the worse.
  The Mini-BESTest consists of 14 tasks that assess static, proactive, and reactive balance. This balance measure is a shorter version of the original 27-item BESTest and takes only 15 minutes to administer. The mini-BESTest may be more appropriate and effective for ambulatory people with MS with relatively few walking disabilities. Higher scores mean better outcome.
V3 visit- Mini-BESTest | 9 months after V0 visit
  Mini-BESTest - Balance Evaluation Systems Test measure in points from 0 - 28. Objective test (clinical), The less, the worse.
  The Mini-BESTest consists of 14 tasks that assess static, proactive, and reactive balance. This balance measure is a shorter version of the original 27-item BESTest and takes only 15 minutes to administer. The mini-BESTest may be more appropriate and effective for ambulatory people with MS with relatively few walking disabilities. Higher scores mean better outcome.
V4 visit- Mini-BESTest | 12 months after V0 visit
  Mini-BESTest - Balance Evaluation Systems Test measure in points from 0 - 28. Objective test (clinical), The less, the worse.
  The Mini-BESTest consists of 14 tasks that assess static, proactive, and reactive balance. This balance measure is a shorter version of the original 27-item BESTest and takes only 15 minutes to administer. The mini-BESTest may be more appropriate and effective for ambulatory people with MS with relatively few walking disabilities. Higher scores mean better outcome.

SECONDARY OUTCOMES:
V0 visit- EDSS - Expanded disability status scale | 1. day
  EDSS - Expanded disability status scale in points from 0 - 10, Ordinal rating system, The more, the worse
V1 visit- EDSS - Expanded disability status scale | 3 months after V0 visit
  EDSS - Expanded disability status scale in points from 0 - 10, Ordinal rating system, The more, the worse
V2 visit- EDSS - Expanded disability status scale | 6 months after V0 visit
  EDSS - Expanded disability status scale in points from 0 - 10, Ordinal rating system, The more, the worse
V3 visit- EDSS - Expanded disability status scale | 9 months after V0 visit
  EDSS - Expanded disability status scale in points from 0 - 10, Ordinal rating system, The more, the worse
V4 visit- EDSS - Expanded disability status scale | 12 months after V0 visit
  EDSS - Expanded disability status scale in points from 0 - 10, Ordinal rating system, The more, the worse
V0 visit- T25FW - Timed 25-foot walk test | 1. day
  T25FW - Timed 25-foot walk test in seconds, Objective test (clinical), The more, the worse.
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score for the T25-FW is the average of the two completed trials. Higher scores mean worse outcome.
V1 visit- T25FW - Timed 25-foot walk test | 3 months after V0 visit
  T25FW - Timed 25-foot walk test in seconds, Objective test (clinical), The more, the worse.
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score for the T25-FW is the average of the two completed trials. Higher scores mean worse outcome.
V2 visit- T25FW - Timed 25-foot walk test | 6 months after V0 visit
  T25FW - Timed 25-foot walk test in seconds, Objective test (clinical), The more, the worse.
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score for the T25-FW is the average of the two completed trials. Higher scores mean worse outcome.
V3 visit- T25FW - Timed 25-foot walk test | 9 months after V0 visit
  T25FW - Timed 25-foot walk test in seconds, Objective test (clinical), The more, the worse.
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score for the T25-FW is the average of the two completed trials. Higher scores mean worse outcome.
V4 visit- T25FW - Timed 25-foot walk test | 12 months after V0 visit
  T25FW - Timed 25-foot walk test in seconds, Objective test (clinical), The more, the worse.
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task. The score for the T25-FW is the average of the two completed trials. Higher scores mean worse outcome.
V0 visit- PASAT - Paced Auditory Serial Addition | 1. day
  PASAT - Paced Auditory Serial Addition in correct items from 0 - 60, Scale, The less, the worse.
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. The PASAT is presented using audio cassette tape or compact disk to ensure standardization in the rate of stimulus presentation. The score for the PASAT is the total number correct out of 60 possible answers. Higher scores mean better outcome.
V1 visit- PASAT - Paced Auditory Serial Addition | 3 months after V0 visit
  PASAT - Paced Auditory Serial Addition in correct items from 0 - 60, Scale, The less, the worse.
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. The PASAT is presented using audio cassette tape or compact disk to ensure standardization in the rate of stimulus presentation. The score for the PASAT is the total number correct out of 60 possible answers. Higher scores mean better outcome.
V2 visit- PASAT - Paced Auditory Serial Addition | 6 months after V0 visit
  PASAT - Paced Auditory Serial Addition in correct items from 0 - 60, Scale, The less, the worse.
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. The PASAT is presented using audio cassette tape or compact disk to ensure standardization in the rate of stimulus presentation. The score for the PASAT is the total number correct out of 60 possible answers. Higher scores mean better outcome.
V3 visit- PASAT - Paced Auditory Serial Addition | 9 months after V0 visit
  PASAT - Paced Auditory Serial Addition in correct items from 0 - 60, Scale, The less, the worse.
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. The PASAT is presented using audio cassette tape or compact disk to ensure standardization in the rate of stimulus presentation. The score for the PASAT is the total number correct out of 60 possible answers. Higher scores mean better outcome.
V4 visit- PASAT - Paced Auditory Serial Addition | 12 months after V0 visit
  PASAT - Paced Auditory Serial Addition in correct items from 0 - 60, Scale, The less, the worse.
  The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. The PASAT is presented using audio cassette tape or compact disk to ensure standardization in the rate of stimulus presentation. The score for the PASAT is the total number correct out of 60 possible answers. Higher scores mean better outcome.
V0 visit- SDMT - Symbol Digit Modalities Test | 1. day
  SDMT - Symbol Digit Modalities Test in correct items from 0 - 110, Scale, The less, the worse.
  The Symbol Digit Modalities Test (SDMT) is the most sensitive screening metric of neurocognitive function in multiple sclerosis (MS) and is consistently interpreted as a measure of information processing speed (IPS), attention and working memory. It is a paper-pencil measure which requires an individual to substitute digits for abstract symbols using a reference key. Higher scores mean better outcome.
V1 visit- SDMT - Symbol Digit Modalities Test | 3 months after V0 visit
  SDMT - Symbol Digit Modalities Test in correct items from 0 - 110, Scale, The less, the worse.
  The Symbol Digit Modalities Test (SDMT) is the most sensitive screening metric of neurocognitive function in multiple sclerosis (MS) and is consistently interpreted as a measure of information processing speed (IPS), attention and working memory. It is a paper-pencil measure which requires an individual to substitute digits for abstract symbols using a reference key. Higher scores mean better outcome.
V2 visit- SDMT - Symbol Digit Modalities Test | 6 months after V0 visit
  SDMT - Symbol Digit Modalities Test in correct items from 0 - 110, Scale, The less, the worse.
  The Symbol Digit Modalities Test (SDMT) is the most sensitive screening metric of neurocognitive function in multiple sclerosis (MS) and is consistently interpreted as a measure of information processing speed (IPS), attention and working memory. It is a paper-pencil measure which requires an individual to substitute digits for abstract symbols using a reference key. Higher scores mean better outcome.
V3 visit- SDMT - Symbol Digit Modalities Test | 9 months after V0 visit
  SDMT - Symbol Digit Modalities Test in correct items from 0 - 110, Scale, The less, the worse.
  The Symbol Digit Modalities Test (SDMT) is the most sensitive screening metric of neurocognitive function in multiple sclerosis (MS) and is consistently interpreted as a measure of information processing speed (IPS), attention and working memory. It is a paper-pencil measure which requires an individual to substitute digits for abstract symbols using a reference key. Higher scores mean better outcome.
V4 visit- SDMT - Symbol Digit Modalities Test | 12 months after V0 visit
  SDMT - Symbol Digit Modalities Test in correct items from 0 - 110, Scale, The less, the worse.
  The Symbol Digit Modalities Test (SDMT) is the most sensitive screening metric of neurocognitive function in multiple sclerosis (MS) and is consistently interpreted as a measure of information processing speed (IPS), attention and working memory. It is a paper-pencil measure which requires an individual to substitute digits for abstract symbols using a reference key. Higher scores mean better outcome.
V0 visit- EQ-5D - European Quality of Life Questionnaire | 1. day
  The EQ-5D is a measure of self-reported health outcomes that is applicable to a wide range of health conditions and treatments. It consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II). Part I of the scale consists of 5 single-item dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a 3 point response scale designed to indicate the level of the problem. Part II uses a vertical graduated VAS (thermometer) to measure health status, ranging from worst imaginable health state to best imaginable health state. Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Higher scores mean worse outcome. Part II is scored from 0 to 100. The score from Part II can be used to track changes in health, on an individual or group level, over time. Higher scores mean better outcome.
V1 visit- EQ-5D - European Quality of Life Questionnaire | 3 months after V0 visit
  The EQ-5D is a measure of self-reported health outcomes that is applicable to a wide range of health conditions and treatments. It consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II). Part I of the scale consists of 5 single-item dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a 3 point response scale designed to indicate the level of the problem. Part II uses a vertical graduated VAS (thermometer) to measure health status, ranging from worst imaginable health state to best imaginable health state. Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Higher scores mean worse outcome. Part II is scored from 0 to 100. The score from Part II can be used to track changes in health, on an individual or group level, over time. Higher scores mean better outcome.
V2 visit- EQ-5D - European Quality of Life Questionnaire | 6 months after V0 visit
  The EQ-5D is a measure of self-reported health outcomes that is applicable to a wide range of health conditions and treatments. It consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II). Part I of the scale consists of 5 single-item dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a 3 point response scale designed to indicate the level of the problem. Part II uses a vertical graduated VAS (thermometer) to measure health status, ranging from worst imaginable health state to best imaginable health state. Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Higher scores mean worse outcome. Part II is scored from 0 to 100. The score from Part II can be used to track changes in health, on an individual or group level, over time. Higher scores mean better outcome.
V3 visit- EQ-5D - European Quality of Life Questionnaire | 9 months after V0 visit
  The EQ-5D is a measure of self-reported health outcomes that is applicable to a wide range of health conditions and treatments. It consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II). Part I of the scale consists of 5 single-item dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a 3 point response scale designed to indicate the level of the problem. Part II uses a vertical graduated VAS (thermometer) to measure health status, ranging from worst imaginable health state to best imaginable health state. Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Higher scores mean worse outcome. Part II is scored from 0 to 100. The score from Part II can be used to track changes in health, on an individual or group level, over time. Higher scores mean better outcome.
V4 visit- EQ-5D - European Quality of Life Questionnaire | 12 months after V0 visit
  The EQ-5D is a measure of self-reported health outcomes that is applicable to a wide range of health conditions and treatments. It consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II). Part I of the scale consists of 5 single-item dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a 3 point response scale designed to indicate the level of the problem. Part II uses a vertical graduated VAS (thermometer) to measure health status, ranging from worst imaginable health state to best imaginable health state. Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Higher scores mean worse outcome. Part II is scored from 0 to 100. The score from Part II can be used to track changes in health, on an individual or group level, over time. Higher scores mean better outcome.
V0 visit- FES - Falls Efficacy Scale | 1. day
  FES - Falls Efficacy Scale in points from 0 - 100, Questionnaire, The more, the worse The FES is a questionnaire assessing the confidence level individuals have in performing daily activities without falling. The FES is a 10 item scale where each item is rated on a scale of 1-10. A score of 10 signifies no confidence in these activities; a score of 1 indicates confidence. Higher scores mean worse outcome. Out of a total score of 100, a score of 70 or above indicates the individual has a fear of falling.
V1 visit- FES - Falls Efficacy Scale | 3 months after V0 visit
  FES - Falls Efficacy Scale in points from 0 - 100, Questionnaire, The more, the worse The FES is a questionnaire assessing the confidence level individuals have in performing daily activities without falling. The FES is a 10 item scale where each item is rated on a scale of 1-10. A score of 10 signifies no confidence in these activities; a score of 1 indicates confidence. Higher scores mean worse outcome. Out of a total score of 100, a score of 70 or above indicates the individual has a fear of falling.
V2 visit- FES - Falls Efficacy Scale | 6 months after V0 visit
  FES - Falls Efficacy Scale in points from 0 - 100, Questionnaire, The more, the worse The FES is a questionnaire assessing the confidence level individuals have in performing daily activities without falling. The FES is a 10 item scale where each item is rated on a scale of 1-10. A score of 10 signifies no confidence in these activities; a score of 1 indicates confidence. Higher scores mean worse outcome. Out of a total score of 100, a score of 70 or above indicates the individual has a fear of falling.
V3 visit- FES - Falls Efficacy Scale | 9 months after V0 visit
  FES - Falls Efficacy Scale in points from 0 - 100, Questionnaire, The more, the worse The FES is a questionnaire assessing the confidence level individuals have in performing daily activities without falling. The FES is a 10 item scale where each item is rated on a scale of 1-10. A score of 10 signifies no confidence in these activities; a score of 1 indicates confidence. Higher scores mean worse outcome. Out of a total score of 100, a score of 70 or above indicates the individual has a fear of falling.
V4 visit- FES - Falls Efficacy Scale | 12 months after V0 visit
  FES - Falls Efficacy Scale in points from 0 - 100, Questionnaire, The more, the worse The FES is a questionnaire assessing the confidence level individuals have in performing daily activities without falling. The FES is a 10 item scale where each item is rated on a scale of 1-10. A score of 10 signifies no confidence in these activities; a score of 1 indicates confidence. Higher scores mean worse outcome. Out of a total score of 100, a score of 70 or above indicates the individual has a fear of falling.
V0 visit- ABC - Activities-Specific Balance Confidence Scale | 1. day
  ABC - Activities-Specific Balance Confidence Scale in points from 0 - 150, Questionnaire, The less, the worse Perceived balance confidence was evaluated by Activity Balance Confidence scale (ABC). This test assesses the self-reported patient´s level of confidence while performing a continuum of less and more challenging 16 common daily activities. Higher scores mean better outcome. A score of > 80% indicates high level of functioning
V1 visit- ABC - Activities-Specific Balance Confidence Scale | 3 months after V0 visit
  ABC - Activities-Specific Balance Confidence Scale in points from 0 - 150, Questionnaire, The less, the worse Perceived balance confidence was evaluated by Activity Balance Confidence scale (ABC). This test assesses the self-reported patient´s level of confidence while performing a continuum of less and more challenging 16 common daily activities. Higher scores mean better outcome. A score of > 80% indicates high level of functioning
V2 visit- ABC - Activities-Specific Balance Confidence Scale | 6 months after V0 visit
  ABC - Activities-Specific Balance Confidence Scale in points from 0 - 150, Questionnaire, The less, the worse Perceived balance confidence was evaluated by Activity Balance Confidence scale (ABC). This test assesses the self-reported patient´s level of confidence while performing a continuum of less and more challenging 16 common daily activities. Higher scores mean better outcome. A score of > 80% indicates high level of functioning
V3 visit- ABC - Activities-Specific Balance Confidence Scale | 9 months after V0 visit
  ABC - Activities-Specific Balance Confidence Scale in points from 0 - 150, Questionnaire, The less, the worse Perceived balance confidence was evaluated by Activity Balance Confidence scale (ABC). This test assesses the self-reported patient´s level of confidence while performing a continuum of less and more challenging 16 common daily activities. Higher scores mean better outcome. A score of > 80% indicates high level of functioning
V4 visit- ABC - Activities-Specific Balance Confidence Scale | 12 months after V0 visit
  ABC - Activities-Specific Balance Confidence Scale in points from 0 - 150, Questionnaire, The less, the worse Perceived balance confidence was evaluated by Activity Balance Confidence scale (ABC). This test assesses the self-reported patient´s level of confidence while performing a continuum of less and more challenging 16 common daily activities. Higher scores mean better outcome. A score of > 80% indicates high level of functioning
V0 visit- BDI-II - The Beck Depression Inventory | 1. day
  BDI-II - The Beck Depression Inventory in points from 0 - 63, Questionnaire, The more, the worse The Beck Depression Inventory (BDI-II) is a widely clinically used 21-item self-reported scale to evaluate the severity of depression. The Beck Anxiety Inventory (BAI) is self-reported 21-scale to evaluate the level of anxiety. Both of scales minimum value is 0 and maximum value is 63. Higher scores mean worse outcome
V1 visit- BDI-II - The Beck Depression Inventory | 3 months after V0 visit
  BDI-II - The Beck Depression Inventory in points from 0 - 63, Questionnaire, The more, the worse The Beck Depression Inventory (BDI-II) is a widely clinically used 21-item self-reported scale to evaluate the severity of depression. The Beck Anxiety Inventory (BAI) is self-reported 21-scale to evaluate the level of anxiety. Both of scales minimum value is 0 and maximum value is 63. Higher scores mean worse outcome
V2 visit- BDI-II - The Beck Depression Inventory | 6 months after V0 visit
  BDI-II - The Beck Depression Inventory in points from 0 - 63, Questionnaire, The more, the worse The Beck Depression Inventory (BDI-II) is a widely clinically used 21-item self-reported scale to evaluate the severity of depression. The Beck Anxiety Inventory (BAI) is self-reported 21-scale to evaluate the level of anxiety. Both of scales minimum value is 0 and maximum value is 63. Higher scores mean worse outcome
V3 visit- BDI-II - The Beck Depression Inventory | 9 months after V0 visit
  BDI-II - The Beck Depression Inventory in points from 0 - 63, Questionnaire, The more, the worse The Beck Depression Inventory (BDI-II) is a widely clinically used 21-item self-reported scale to evaluate the severity of depression. The Beck Anxiety Inventory (BAI) is self-reported 21-scale to evaluate the level of anxiety. Both of scales minimum value is 0 and maximum value is 63. Higher scores mean worse outcome
V4 visit- BDI-II - The Beck Depression Inventory | 12 months after V0 visit
  BDI-II - The Beck Depression Inventory in points from 0 - 63, Questionnaire, The more, the worse The Beck Depression Inventory (BDI-II) is a widely clinically used 21-item self-reported scale to evaluate the severity of depression. The Beck Anxiety Inventory (BAI) is self-reported 21-scale to evaluate the level of anxiety. Both of scales minimum value is 0 and maximum value is 63. Higher scores mean worse outcome
V0 visit- BAI - The Beck Anxiety Inventory | 1. day
  BAI - The Beck Anxiety Inventory in points from 0 - 63, Questionnaire, The more, the worse
V1 visit- BAI - The Beck Anxiety Inventory | 3 months after V0 visit
  BAI - The Beck Anxiety Inventory in points from 0 - 63, Questionnaire, The more, the worse
V2 visit- BAI - The Beck Anxiety Inventory | 6 months after V0 visit
  BAI - The Beck Anxiety Inventory in points from 0 - 63, Questionnaire, The more, the worse
V3 visit- BAI - The Beck Anxiety Inventory | 9 months after V0 visit
  BAI - The Beck Anxiety Inventory in points from 0 - 63, Questionnaire, The more, the worse
V4 visit- BAI - The Beck Anxiety Inventory | 12 months after V0 visit
  BAI - The Beck Anxiety Inventory in points from 0 - 63, Questionnaire, The more, the worse
V0 visit- MoCA - Montreal cognitive assessment | 1. day
  MoCA - Montreal cognitive assessment in points from 0 - 30, Scale, The less, the worse.
  MoCA is a widely used screening assessment for detecting cognitive impairment. This test consists of 30 points and takes part in 10 minutes from the individual. The Montreal test is performed in seven steps, which may change in some countries dependent on education and culture. The basics of this test include short-term memory, executable performance, attention and focus. Higher scores mean better outcome.
V1 visit- MoCA - Montreal cognitive assessment | 3 months after V0 visit
  MoCA - Montreal cognitive assessment in points from 0 - 30, Scale, The less, the worse.
  MoCA is a widely used screening assessment for detecting cognitive impairment. This test consists of 30 points and takes part in 10 minutes from the individual. The Montreal test is performed in seven steps, which may change in some countries dependent on education and culture. The basics of this test include short-term memory, executable performance, attention and focus. Higher scores mean better outcome.
V2 visit- MoCA - Montreal cognitive assessment | 6 months after V0 visit
  MoCA - Montreal cognitive assessment in points from 0 - 30, Scale, The less, the worse.
  MoCA is a widely used screening assessment for detecting cognitive impairment. This test consists of 30 points and takes part in 10 minutes from the individual. The Montreal test is performed in seven steps, which may change in some countries dependent on education and culture. The basics of this test include short-term memory, executable performance, attention and focus. Higher scores mean better outcome.
V3 visit- MoCA - Montreal cognitive assessment | 9 months after V0 visit
  MoCA - Montreal cognitive assessment in points from 0 - 30, Scale, The less, the worse.
  MoCA is a widely used screening assessment for detecting cognitive impairment. This test consists of 30 points and takes part in 10 minutes from the individual. The Montreal test is performed in seven steps, which may change in some countries dependent on education and culture. The basics of this test include short-term memory, executable performance, attention and focus. Higher scores mean better outcome.
V4 visit- MoCA - Montreal cognitive assessment | 12 months after V0 visit
  MoCA - Montreal cognitive assessment in points from 0 - 30, Scale, The less, the worse.
  MoCA is a widely used screening assessment for detecting cognitive impairment. This test consists of 30 points and takes part in 10 minutes from the individual. The Montreal test is performed in seven steps, which may change in some countries dependent on education and culture. The basics of this test include short-term memory, executable performance, attention and focus. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Valkovič, prof.MD.PhD., Study Chair — 2nd Department of Neurology, Faculty of MedicineCOMENIUS UNIVERSITY BRATISLAVA
Locations (1):
- 2nd Department of Neurology, Faculty of Medicine COMENIUS UNIVERSITY BRATISLAVA, Bratislava, Slovak Republic, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gibson JC, Summers GD. Bone health in multiple sclerosis. Osteoporos Int. 2011 Dec;22(12):2935-49. doi: 10.1007/s00198-011-1644-8. Epub 2011 May 21. PMID 21604009
- [Result] Arnett PA, Strober LB. Cognitive and neurobehavioral features in multiple sclerosis. Expert Rev Neurother. 2011 Mar;11(3):411-24. doi: 10.1586/ern.11.12. PMID 21375446
- [Result] Latimer-Cheung AE, Pilutti LA, Hicks AL, Martin Ginis KA, Fenuta AM, MacKibbon KA, Motl RW. Effects of exercise training on fitness, mobility, fatigue, and health-related quality of life among adults with multiple sclerosis: a systematic review to inform guideline development. Arch Phys Med Rehabil. 2013 Sep;94(9):1800-1828.e3. doi: 10.1016/j.apmr.2013.04.020. Epub 2013 May 10. PMID 23669008
- [Result] Alvarenga-Filho H, Sacramento PM, Ferreira TB, Hygino J, Abreu JEC, Carvalho SR, Wing AC, Alvarenga RMP, Bento CAM. Combined exercise training reduces fatigue and modulates the cytokine profile of T-cells from multiple sclerosis patients in response to neuromediators. J Neuroimmunol. 2016 Apr 15;293:91-99. doi: 10.1016/j.jneuroim.2016.02.014. Epub 2016 Feb 26. PMID 27049568
- [Result] Wens I, Keytsman C, Deckx N, Cools N, Dalgas U, Eijnde BO. Brain derived neurotrophic factor in multiple sclerosis: effect of 24 weeks endurance and resistance training. Eur J Neurol. 2016 Jun;23(6):1028-35. doi: 10.1111/ene.12976. Epub 2016 Mar 16. PMID 26992038
- [Result] Husted C, Pham L, Hekking A, Niederman R. Improving quality of life for people with chronic conditions: the example of t'ai chi and multiple sclerosis. Altern Ther Health Med. 1999 Sep;5(5):70-4. PMID 10484833
- [Result] Azimzadeh E, Hosseini MA, Nourozi K, Davidson PM. Effect of Tai Chi Chuan on balance in women with multiple sclerosis. Complement Ther Clin Pract. 2015 Feb;21(1):57-60. doi: 10.1016/j.ctcp.2014.09.002. Epub 2014 Nov 27. PMID 25534298
- [Result] Burschka JM, Keune PM, Oy UH, Oschmann P, Kuhn P. Mindfulness-based interventions in multiple sclerosis: beneficial effects of Tai Chi on balance, coordination, fatigue and depression. BMC Neurol. 2014 Aug 23;14:165. doi: 10.1186/s12883-014-0165-4. PMID 25145392
- [Derived] Menkyova I, Stastna D, Novotna K, Saling M, Lisa I, Vesely T, Slezakova D, Valkovic P. Effect of Tai-chi on balance, mood, cognition, and quality of life in women with multiple sclerosis: A one-year prospective study. Explore (NY). 2024 Mar-Apr;20(2):188-195. doi: 10.1016/j.explore.2023.07.011. Epub 2023 Aug 6. PMID 37596158